CLINICAL TRIAL: NCT01896037
Title: Omega-3 Supplementation to Increase HDL-c Levels in Those With Tetraplegia
Brief Title: Omega-3 Supplementation for Tetraplegics With Poor Cholesterol Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: The Association of Rehabilitation Medicine in Manitoba (Unknown)
Responsible Party: Principal Investigator, Dr. Karen Ethans, Director, Spinal Cord Rehabilitation Unit, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDL2013
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Spinal Cord Injury; Tetraplegia; Quadraplegia; Low HDL-c; High LDL-c
Keywords: Spinal cord injury; Tetraplegia; Quadraplegia; Cholesterol; HDL-c; LDL-c; Omega-3 fatty acids
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega-3 supplements (Experimental): Daily omega-3 supplements of 600 mg EPA (Eicosapentaenoic acid) and 300 mg DHA (Docosahexaenoic acid) for 5 months.
  Interventions: Dietary Supplement: Omega-3 supplements

INTERVENTIONS:
Dietary Supplement: Omega-3 supplements — Daily omega-3 supplements of 600 mg EPA (Eicosapentaenoic acid) and 300 mg DHA (Docosahexaenoic acid) for 5 months.

SUMMARY:
People with a spinal cord injury (SCI) characteristically have low levels of high-density lipoprotein-cholesterol (HDL-c; "good cholesterol") and high levels of low-density lipoprotein-cholesterol (LDL-c; "bad cholesterol"), and are at a higher risk of developing cardiovascular health problems, such as heart disease, heart attack and stroke, than the able-bodied population. A common way for able-bodied people to improve their lipid profile is through exercise; however, SCI people, especially tetraplegics, are often unable to achieve and maintain a level of exercise needed to obtain these benefits. It is therefore clinically important to find an effective, safe and inexpensive method of increasing HDL-c levels in people with chronic tetraplegia. This study will investigate the effects of omega-3 fatty acid supplementation on the lipid profile of people with tetraplegia. The investigators hypothesize that 5 months of daily consumption of high doses of omega-3 fatty acids will increase plasma levels of HDL-c in those with tetraplegia, leading to decreased risk of cardiovascular health issues.

ELIGIBILITY:
Inclusion Criteria:

* Having chronic tetraplegia (at least on year since injury)
* 18 years or older
* Having below normal fasting blood plasma levels of HDL-c (<1 mmol/l)

Exclusion Criteria:

* Currently taking omega-3 supplements
* Currently taking medications for abnormal cholesterol
* Having a heart attack or stroke in the past one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-01-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
Blood plasma levels of HDL-cholesterol | Month 5
  Change in blood plasma levels of HDL-cholesterol at month 5 compared to baseline levels

SECONDARY OUTCOMES:
Blood plasma levels of total cholesterol | Month 5
  Change in blood plasma levels of total cholesterol at month 5 compared to baseline levels

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ethans, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada